CLINICAL TRIAL: NCT01343004
Title: A Randomized, Double-blind, Placebo-Controlled, Comparative Multicenter Phase 3 Study to Evaluate the Safety and Efficacy of BA058 (Abaloparatide) for Injection for Prevention of Fracture in Ambulatory Postmenopausal Women With Severe Osteoporosis and at Risk of Fracture
Brief Title: Study to Evaluate the Safety and Efficacy of BA058 (Abaloparatide) for Prevention of Fracture in Postmenopausal Women
Acronym: ACTIVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radius Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BA058-05-003; ACTIVE Trial (Other: Radius Health, Inc.)
Record Dates: First submitted 2011-04-26; First posted 2011-04-27 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-01

CONDITIONS: Osteoporosis; Postmenopausal Osteoporosis
Keywords: BA058; abaloparatide; Abaloparatide-SC; osteoporosis; postmenopausal; bone loss; ACTIVE; fracture
MeSH Terms: conditions — Osteoporosis; Osteoporosis, Postmenopausal; Bone Diseases, Metabolic; Motor Activity; Fractures, Bone | interventions — abaloparatide; Teriparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo identical in appearance to BA058 study drug
  Interventions: Drug: Placebo
- BA058 80 mcg (abaloparatide) (Experimental)
  Interventions: Drug: BA058 80 mcg
- teriparatide (Active Comparator): Blinded until after randomization, then open-label
  Interventions: Drug: teriparatide

INTERVENTIONS:
Drug: Placebo — Placebo 0 mcg subcutaneous daily
  Arms: Placebo
Drug: BA058 80 mcg — BA058 80 mcg subcutaneous daily
  Other Names: abaloparatide, Abaloparatide-SC
  Arms: BA058 80 mcg (abaloparatide)
Drug: teriparatide — teriparatide 20 mcg subcutaneous daily
  Other Names: Forteo; Forsteo
  Arms: teriparatide

SUMMARY:
The purpose of this study is to determine whether BA058 (abaloparatide), a parathyroid hormone-related peptide, is effective in preventing fractures in postmenopausal women with severe osteoporosis who are at risk of fractures.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, comparative Phase 3, multicenter international study to evaluate the efficacy and safety of BA058 (abaloparatide) 80 µg in the prevention of fracture in otherwise healthy ambulatory postmenopausal women with severe osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy ambulatory postmenopausal (≥ 5 years) women from 50 to 85 years of age (inclusive) with a diagnosis of osteoporosis
* The women are to have a bone mineral density (BMD) T score ≤ -2.5 and > -5.0 at the lumbar spine or hip (femoral neck) by dual energy x-ray absorptiometry (DXA) and radiological evidence of 2 or more mild or one or more moderate lumbar or thoracic vertebral fractures, or history of low trauma forearm, humerus, sacral, pelvic, hip, femoral, or tibial fracture within the past 5 years. Postmenopausal women older than 65 who meet the above fracture criteria but have a T score ≤ -2.0 and > -5.0 may be enrolled. Women older than 65 who do not meet the fracture criteria may also be enrolled if their T score is ≤ -3.0 and > -5.0
* Normal physical exam, vital signs, electrocardiogram (ECG) and medical history
* Laboratory tests within the normal range including serum calcium, PTH(1-84), serum phosphorus and alkaline phosphatase

Exclusion Criteria:

* History of more than 4 mild or moderate spine fractures or any severe fracture
* Abnormality of the spine or hip that would prohibit assessment of bone mineral density (BMD)
* Unexplained elevation of serum alkaline phosphatase, history of bone disorders (such as Paget's disease) or a diagnosis of cancer within the last 5 years (with the exception of basal cell or squamous cancer of the skin)
* History of thyroid, parathyroid, or adrenal disorders, or malabsorptive syndromes or any chronic or recurrent diseases or disturbances that would interfere with the interpretation of study data or compromise the safety of the patient
* Prior treatment with parathyroid hormone (PTH) or parathyroid hormone-related peptid (PTHrP)
* Prior treatment with bisphosphonates, fluoride, or strontium within the past five years or treatment with androgens, anabolic steroids, corticosteroids or selective estrogen receptor modulators within the past 12 months (except hormone replacement therapy)
* Prior treatment with an investigational drug within the past 12 months
* History of nephrolithiasis or urolithiasis within the past five years, or history of osteosarcoma at any time

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2463 (Actual)
Dates: Start 2011-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Radius Health, Inc., Study Director — Radius Health, Inc.
Locations (28):
- United States (5):
  - Lakewood, Colorado
  - Miami, Florida
  - North Miami, Florida
  - Atlanta, Georgia
  - Bethesda, Maryland
- Buenos Aires, Argentina
- Brazil (5):
  - Brasília
  - Curitiba
  - Rio de Janeiro
  - São Paulo
  - Vitória
- Czechia (3):
  - Brno
  - Pardubice
  - Prague
- Denmark (3):
  - Aalborg
  - Ballerup Municipality
  - Vejle
- Estonia (2):
  - Tallinn
  - Tartu
- Hong Kong, Hong Kong
- Vilnius, Lithuania
- Poland (6):
  - Bialystok
  - Katowice
  - Kielce
  - Lodz
  - Warsaw
  - Zgierz
- Bucharest, Romania

REFERENCES:
- [Derived] Sheth NP, Krohn K, Torkelson J, Winzenrieth R, Humbert L, Pearman L, Wang Y, Boxberger JI, Bostrom MP. Abaloparatide effects on BMD in acetabular regions corresponding to DeLee and Charnley zones in women with postmenopausal osteoporosis. Bone Rep. 2025 Jul 19;26:101858. doi: 10.1016/j.bonr.2025.101858. eCollection 2025 Sep. PMID 40786602
- [Derived] DeSapri KT, Clarke BL, Kostenuik P, Wang Y, Mitlak BH. Effect of abaloparatide on fracture incidence and bone mineral density in postmenopausal women with osteoporosis at highest risk for fracture. Menopause. 2025 May 1;32(5):388-395. doi: 10.1097/GME.0000000000002516. PMID 39999474
- [Derived] Cosman F, Hans D, Shevroja E, Wang Y, Mitlak B. Effect of Abaloparatide on Bone Microarchitecture Assessed by Trabecular Bone Score in Women With Osteoporosis: Post Hoc Analysis of ACTIVE and ACTIVExtend. J Bone Miner Res. 2023 Apr;38(4):464-470. doi: 10.1002/jbmr.4764. Epub 2023 Feb 12. PMID 36588166
- [Derived] Hara T, Hijikata Y, Matsubara Y, Watanabe N. Pharmacological interventions versus placebo, no treatment or usual care for osteoporosis in people with chronic kidney disease stages 3-5D. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD013424. doi: 10.1002/14651858.CD013424.pub2. PMID 34231877
- [Derived] Cosman F, Peterson LR, Towler DA, Mitlak B, Wang Y, Cummings SR. Cardiovascular Safety of Abaloparatide in Postmenopausal Women With Osteoporosis: Analysis From the ACTIVE Phase 3 Trial. J Clin Endocrinol Metab. 2020 Nov 1;105(11):3384-95. doi: 10.1210/clinem/dgaa450. PMID 32658264
- [Derived] Saag KG, Williams SA, Wang Y, Weiss RJ, Cauley JA. Effect of Abaloparatide on Bone Mineral Density and Fracture Incidence in a Subset of Younger Postmenopausal Women with Osteoporosis at High Risk for Fracture. Clin Ther. 2020 Jun;42(6):1099-1107.e1. doi: 10.1016/j.clinthera.2020.04.012. Epub 2020 Jun 6. PMID 32513495
- [Derived] Leder BZ, Mitlak B, Hu MY, Hattersley G, Bockman RS. Effect of Abaloparatide vs Alendronate on Fracture Risk Reduction in Postmenopausal Women With Osteoporosis. J Clin Endocrinol Metab. 2020 Mar 1;105(3):938-43. doi: 10.1210/clinem/dgz162. PMID 31674644
- [Derived] Leder BZ, Zapalowski C, Hu MY, Hattersley G, Lane NE, Singer AJ, Dore RK. Fracture and Bone Mineral Density Response by Baseline Risk in Patients Treated With Abaloparatide Followed by Alendronate: Results From the Phase 3 ACTIVExtend Trial. J Bone Miner Res. 2019 Dec;34(12):2213-2219. doi: 10.1002/jbmr.3848. Epub 2019 Sep 11. PMID 31411768
- [Derived] Moreira CA, Fitzpatrick LA, Wang Y, Recker RR. Effects of abaloparatide-SC (BA058) on bone histology and histomorphometry: The ACTIVE phase 3 trial. Bone. 2017 Apr;97:314-319. doi: 10.1016/j.bone.2016.11.004. Epub 2016 Nov 5. PMID 27826127
- [Derived] Cosman F, Hattersley G, Hu MY, Williams GC, Fitzpatrick LA, Black DM. Effects of Abaloparatide-SC on Fractures and Bone Mineral Density in Subgroups of Postmenopausal Women With Osteoporosis and Varying Baseline Risk Factors. J Bone Miner Res. 2017 Jan;32(1):17-23. doi: 10.1002/jbmr.2991. Epub 2016 Sep 28. PMID 27612281
- [Derived] Miller PD, Hattersley G, Riis BJ, Williams GC, Lau E, Russo LA, Alexandersen P, Zerbini CA, Hu MY, Harris AG, Fitzpatrick LA, Cosman F, Christiansen C; ACTIVE Study Investigators. Effect of Abaloparatide vs Placebo on New Vertebral Fractures in Postmenopausal Women With Osteoporosis: A Randomized Clinical Trial. JAMA. 2016 Aug 16;316(7):722-33. doi: 10.1001/jama.2016.11136. PMID 27533157

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | BA058 80 mcg (Abaloparatide) | Teriparatide
Started | 821 | 824 | 818
Completed | 637 | 606 | 658
Not Completed | 184 | 218 | 160

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population included all patients who were randomized into the study by assigning the randomized study medication kit on Day 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BA058 80 mcg (Abaloparatide) | Teriparatide | Total
Number analyzed (Participants) | 821 | 824 | 818 | 2463
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (6.5) | 68.9 (6.5) | 68.8 (6.6) | 68.8 (6.5)
Gender [Count of Participants; unit: Participants]
  Female | 821 | 824 | 818 | 2463
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With New Vertebral Fractures at 18 Months
Time Frame: 18 months
Population: Modified intent-to-treat (MITT) population included all patients with pre-treatment and end-of-treatment evaluable radiologic assessment (spine X-ray).
Measure: Number; unit: participants
Arm/Group | Placebo | BA058 80 mcg (Abaloparatide) | Teriparatide
Number analyzed (Participants) | 711 | 690 | 717
participants | 30 | 4 | 6
Statistical Analysis 1: Comparison: Placebo vs BA058 80 mcg (Abaloparatide); Test type: Superiority or Other; p < 0.0001, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs Teriparatide; Test type: Superiority or Other; p < 0.0001, Fisher Exact

2. Secondary Outcome: Percent Change in Bone Mineral Density (BMD) of Lumbar Spine From Baseline to 18 Months
Time Frame: Basline and 18 months
Population: Intent-to-treat population included all patients who were randomized into the study by assigning the randomized study medication kit on Day 1. Baseline BMD data were missing for some patients; the method of last observation carried forward (LOCF) was used to impute missing data.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Placebo | BA058 80 mcg (Abaloparatide) | Teriparatide
Number analyzed (Participants) | 821 | 823 | 818
percent change from baseline | 0.48 (3.82) | 9.20 (7.54) | 9.12 (6.28)
Statistical Analysis 1: Comparison: Placebo vs BA058 80 mcg (Abaloparatide); Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values were derived from contrast tests based on the ANCOVA model fitted using only the data of the two treatment groups to be compared
Statistical Analysis 2: Comparison: Placebo vs Teriparatide; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: BA058 80 mcg (Abaloparatide) vs Teriparatide; Test type: Superiority or Other; p = 0.8155, ANCOVA; [statistical method as in outcome 2, analysis 1]

3. Secondary Outcome: Percent Change in Bone Mineral Density (BMD) of Total Hip From Baseline to Month 18
Time Frame: Baseline and 18 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | BA058 80 mcg (Abaloparatide) | Teriparatide
Number analyzed (Participants) | 820 | 822 | 818
percent change | -0.08 (2.77) | 3.44 (3.51) | 2.81 (3.33)
Statistical Analysis 1: Comparison: Placebo vs BA058 80 mcg (Abaloparatide); Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Teriparatide; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: BA058 80 mcg (Abaloparatide) vs Teriparatide; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]

4. Secondary Outcome: Percent Change in Bone Mineral Density (BMD) of Femoral Neck From Baseline to Month 18
Time Frame: Baseline and 18 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | BA058 80 mcg (Abaloparatide) | Teriparatide
Number analyzed (Participants) | 820 | 822 | 818
percent change | -0.44 (3.57) | 2.90 (4.21) | 2.26 (3.57)
Statistical Analysis 1: Comparison: Placebo vs BA058 80 mcg (Abaloparatide); Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Teriparatide; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: BA058 80 mcg (Abaloparatide) vs Teriparatide; Test type: Superiority or Other; p = 0.0004, ANCOVA; [statistical method as in outcome 2, analysis 1]

5. Secondary Outcome: Number of Participants With Non-vertebral Fractures at 18 Months
Time Frame: 18 months
Population: Intent-to-treat population included all patients who were randomized into the study by assigning the randomized study medication kit on Day 1.
Measure: Number; unit: Participants
Arm/Group | Placebo | BA058 80 mcg (Abaloparatide) | Teriparatide
Number analyzed (Participants) | 821 | 824 | 818
Participants | 33 | 18 | 24
Statistical Analysis 1: Comparison: Placebo vs BA058 80 mcg (Abaloparatide); Test type: Superiority or Other; p = 0.0318, Chi-squared
Statistical Analysis 2: Comparison: Placebo vs Teriparatide; Test type: Superiority or Other; p = 0.2304, Chi-squared
Statistical Analysis 3: Comparison: BA058 80 mcg (Abaloparatide) vs Teriparatide; Test type: Superiority or Other; p = 0.3361, Chi-squared

6. Secondary Outcome: Number of Treatment-Emergent Adverse Events Associated With Hypercalcemia at 18 Months
Time Frame: 18 months
Population: Safety population included all patients who received 1 or more doses of study medication
Measure: Number; unit: Hypercalcemic events
Arm/Group | Placebo | BA058 80 mcg (Abaloparatide) | Teriparatide
Number analyzed (Participants) | 820 | 822 | 818
Hypercalcemic events | 5 | 15 | 34

ADVERSE EVENTS:
Arm/Group | Placebo | BA058 80 mcg (Abaloparatide) | Teriparatide
Serious Adverse Events (participants affected / at risk) | 90/820 | 80/822 | 82/818
Other Adverse Events (participants affected / at risk) | 447/820 | 492/822 | 456/818
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=820) | BA058 80 mcg (Abaloparatide) (N=822) | Teriparatide (N=818)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 2 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 2 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 1
Myocardial infraction (Cardiac disorders) | 2 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0
Mitral valve stenosis (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 1
Goitre (Endocrine disorders) | 1 | 1 | 2
Thyroid cyst (Endocrine disorders) | 0 | 0 | 1
Malculopathy (Eye disorders) | 0 | 1 | 0
Retinal artery occulusion (Eye disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 2 | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 0 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Change of bowel habit (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 1
Enterocele (Gastrointestinal disorders) | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 2 | 0 | 0
Chest pain (General disorders) | 2 | 1 | 1
Pyrexia (General disorders) | 1 | 1 | 0
Chest discomfort (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1
Sudden death (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 3 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 1
Sepsis (Infections and infestations) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 1
Bronchiolitis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1
Bacterial infection (Infections and infestations) | 1 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Helicobacter infection (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Paronychia (Infections and infestations) | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Postoperative hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 3 | 0 | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Weight decreased (Investigations) | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1
Body temperature increased (Investigations) | 0 | 0 | 1
Bronchoscopy (Investigations) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lumbar spine stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spondylisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 6
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Angiolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bile duct adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Chronic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 2 | 2
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 0
Radicular syndrome (Nervous system disorders) | 0 | 1 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0
Subarchnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 2
Ischaemic stroke (Nervous system disorders) | 3 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 2 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 2 | 0
Uterine prolapse (Reproductive system and breast disorders) | 2 | 2 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 3
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermititis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 1 | 0
Colporrhaphy (Surgical and medical procedures) | 1 | 1 | 0
Coronary angioplasty (Surgical and medical procedures) | 0 | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 1 | 0
Joint arthroplasty (Surgical and medical procedures) | 0 | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 1 | 0 | 1
Osteosynthesis (Surgical and medical procedures) | 0 | 0 | 1
Rectocele repair (Surgical and medical procedures) | 1 | 0 | 0
Removal of internal fixation (Surgical and medical procedures) | 1 | 0 | 0
Toe operation (Surgical and medical procedures) | 0 | 0 | 1
Intermittent claudication (Vascular disorders) | 0 | 1 | 1
Aortic dissection (Vascular disorders) | 1 | 0 | 1
Essential hypertension (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 2
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=820) | BA058 80 mcg (Abaloparatide) (N=822) | Teriparatide (N=818)
Palpitations (Cardiac disorders) | 3 | 42 | 13
Constipation (Gastrointestinal disorders) | 42 | 36 | 34
Nausea (Gastrointestinal disorders) | 25 | 68 | 42
Influenza (Infections and infestations) | 39 | 52 | 34
Nasopharyngitis (Infections and infestations) | 66 | 48 | 52
Upper respiratory tract infection (Infections and infestations) | 63 | 68 | 73
Urinary tract infection (Infections and infestations) | 38 | 43 | 41
Arthralgia (Musculoskeletal and connective tissue disorders) | 80 | 71 | 70
Back pain (Musculoskeletal and connective tissue disorders) | 81 | 69 | 58
Pain in extremity (Musculoskeletal and connective tissue disorders) | 49 | 40 | 42
Hypercalciuria (Renal and urinary disorders) | 74 | 93 | 102
Hypertension (Vascular disorders) | 52 | 59 | 41
Dizziness (Nervous system disorders) | 50 | 82 | 59
Headache (Nervous system disorders) | 49 | 62 | 51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results may not be published prior to the Study Report completion. Investigators may publish results, providing a manuscript to the Sponsor =/> 30 days prior to its submission to a publisher. Sponsor will provide manuscript to Investigators =/> 30 days prior to its submission. Investigator shall comply with Sponsor's policy, withholding publication for an additional 60 days to permit the Sponsor to obtain patent or other proprietary rights protection, if deemed necessary.